CLINICAL TRIAL: NCT04802876
Title: Efficacy of Tislelizumab and Spartalizumab Across Multiple Cancer-types in Patients with PD1-high MRNA Expressing Tumors Defined by a Single and Pre-specified Cutoff
Brief Title: Efficacy of Tislelizumab and Spartalizumab Across Multiple Cancer-types in Patients with PD1-high MRNA Expressing Tumors
Acronym: ACROPOLI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACROPOLI (SOLTI-1904)
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: MSI-H Colorectal Cancer; Melanoma; Anal Carcinoma; Mesothelioma; Triple Negative Breast Cancer; Lung Adenocarcinoma; Cholangiocarcinoma; Cervical Carcinoma; Kidney Clear Cell Carcinoma; Stomach Adenocarcinoma; Esophageal Adenocarcinoma; Uterine Adenocarcinoma; Head and Neck Squamous Cell Carcinoma; Sarcoma; Lung Squamous Cell Carcinoma; Urothelial Carcinoma; Thyroid Carcinoma; Hepatocellular Carcinoma; Uveal Melanoma; HER2-positive Breast Cancer; Pancreatic Adenocarcinoma; Squamous Esophageal Carcinoma; Epithelial Ovarian Cancer; Uterine Carcinosarcoma; Small Cell Lung Cancer; Hormone Receptor Positive / HER2-negative Breast Cancer; Lung Adenocarcinoma EGFR-mutated/ ALK Traslocation; Colorectal Adenocarcinoma; Prostate Adenocarcinoma; Carcinoma of Unknown Primary; Other Histology
Keywords: PD1; Immunotherapy
MeSH Terms: conditions — Melanoma; Anus Neoplasms; Mesothelioma; Triple Negative Breast Neoplasms; Adenocarcinoma of Lung; Cholangiocarcinoma; Uterine Cervical Neoplasms; Carcinoma, Renal Cell; Adenocarcinoma Of Esophagus; Squamous Cell Carcinoma of Head and Neck; Sarcoma; Carcinoma, Transitional Cell; Thyroid Neoplasms; Carcinoma, Hepatocellular; Uveal Melanoma; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Neoplasms, Unknown Primary | interventions — spartalizumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spartalizumab (PDR001) (Cohort-1 PD1-high) (Experimental): 400mg/intravenous every 28 days
  Interventions: Drug: Spartalizumab
- Spartalizumab (PDR001) (Cohort-2 PD1-low) (Experimental): 400mg/intravenous every 28 days
  Interventions: Drug: Spartalizumab
- Tislelizumab (Cohort-3 PD1-high) (Experimental): 300mg/intravenous every 28 days
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Spartalizumab — Spartalizumab (PDR001) 400mg will be given intravenously every 28 days
  Other Names: PDR001
  Arms: Spartalizumab (PDR001) (Cohort-1 PD1-high); Spartalizumab (PDR001) (Cohort-2 PD1-low)
Drug: Tislelizumab — Tislelizumab 300mg will be given intravenously every 28 days
  Arms: Tislelizumab (Cohort-3 PD1-high)

SUMMARY:
This is an open-label, parallel group, non-randomized, multicenter phase II study to evaluate the efficacy of spartalizumab (cohorts 1 and 2) and tislelizumab (cohort 3) in monotherapy in patients with PD1-high-expressing tumors.

DETAILED DESCRIPTION:
Patients will sign a molecular pre-screening consent form across centers in Spain that will allow determination of PD1 mRNA expression on a tumor sample using the nCounter-based technology. This will be centrally performed at Hospital Clinic of Barcelona.

In this trial, three patient cohorts are planned:

* Cohort 1: patients with PD1-high tumors, as defined by the pre-specified cutoff, who will be treated with spartalizumab in monotherapy (400mg/IV every 28 days).
* Cohort 2: patients with PD1-low advanced solid tumors where the efficacy of PD1 / PD-L1 inhibitors has been previously established (i.e. with a FDA or EMA monotherapy indication approved) will also be recruited and treated with spartalizumab in monotherapy (400mg/IV every 28 days).
* Cohort 3: patients with PD1-high tumors, as defined by the pre-specified cutoff, who will be treated with tislelizumab in monotherapy (300mg/IV every 28 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of PD1 mRNA high-expression (cohort 1, 3) or PD1 mRNA low-expression (cohort 2) determined on the tumor sample will be enrolled in this study. Enrollment of patients > 75 years of age is allowed after consultation and approval of the study medical monitor.
2. Life expectancy > 3 months as per investigator opinion.
3. The participant (or legally acceptable representative if applicable) provides written specific informed consent for the remaining screening tests and study procedures before inclusion in the trial.
4. Have measurable disease based on RECIST 1.1 or RANO criteria, as appropriate to tumor type. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Have radiologic evidence of disease progression or recurrence after the previous oncologic treatment
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 10 days prior to the date of allocation.
7. Have adequate organ function. Specimens must be collected within 28 days prior to the start of study treatment.
8. Patients could have received a maximum of 3 lines of prior standard of care chemotherapy in the inoperable/metastatic setting.
9. Treatment-related toxicities (except alopecia) must ≤ Grade 1 at the time of allocation according to CTCAE version 5.0.

Exclusion Criteria:

1. A Women of childbearing potential who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
2. Has received prior therapy with an anti-PD1, anti-PDL1, or anti-PDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
3. Has received prior systemic anti-cancer therapy, including investigational agents within 2 weeks. Medical Monitor could consider shorter interval for kinase inhibitors or other short half-life drugs prior to allocation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline according to CTCAE version 5.0 (except alopecia). Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 2 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 2 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Patients with thymoma are not eligible. Patients with active CNS metastases and/or carcinomatous meningitis are not eligible. Subjects with up to three cerebral metastases are eligible, if all lesions are stable and have been definitively treated with stereotactic radiation therapy, surgery or gamma knife therapy with no evidence of disease progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Has severe hypersensitivity (≥Grade 3) to Spartalizumab or Tislelizumab and/or any of its excipients.
11. History of severe hypersensitivity reactions to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Prior allogeneic stem cell transplantation or organ transplantation
14. Has a history of interstitial lung disease, (non-infectious) pneumonitis that required steroids or has current pneumonitis, uncontrolled lung including pulmonary fibrosis, acute lung diseases, etc. Patients with significantly impaired pulmonary function, or who require supplemental oxygen at baseline must undergo an assessment of pulmonary function at screening.
15. Has an active infection requiring systemic therapy.
16. Has a known history of Human Immunodeficiency Virus (HIV).
17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
18. Has a known history of active TBC (Bacillus Tuberculosis).
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of trial treatment.
22. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 150-days after stopping treatment with spartalizumab or tislelizumab. Highly effective contraception methods include:

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
    4. Placement of a non-hormonal intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year.

    Notes:
    * Double-barrier contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/cream/suppository) are not considered highly effective methods of contraception.
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
23. Sexually active males, unless they use a condom during intercourse while on treatment and for 150 days after stopping treatment with spartalizumab or tislelizumab should not father a child in this period. A condom is required to be used by vasectomized men as well during intercourse in order to prevent delivery of the drug via semen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate (ORR) (Cohort 3) | Until objective tumor response, on average 10 months
  Proportion of patients with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) in patients with high mRNA PD1 expressing tumors (Cohort 3) | Until objective tumor response, on average 10 months
  Proportion of patients with a best overall response of CR, PR or an overall lesion response of Stable Disease (SD) or Non-PR/Non-progression disease (PD) lasting ≥ 24 weeks, based on local investigator´s assessment according to RECIST v1.1.
Progression free survival (PFS) in patients with high mRNA PD1 expressing tumors (Cohort 3) | From date of allocation to disease progression or death from any cause,whichever came first, assessed up to approximately 36 months
  Time from allocation to the first occurrence of disease progression, as determined locally by the investigator using RECIST v.1.1, or death from any cause, whichever occurs first.
Duration of response (DoR) in patients with high mRNA PD1 expressing tumors (Cohort 3) | From date of allocation to disease progression or death from any cause,whichever came first, assessed up to approximately 36 months
  Time from the first occurrence of a documented objective response to disease progression, as determined locally by the investigator through use of RECIST v.1.1, or death from any cause, whichever occurs first
Time to response (TtR) in patients with high mRNA PD1 expressing tumors (Cohort 3) | Until objective tumor response, on average 10 months
  Time from allocation to the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR.
Overall survival (OS) in patients with high mRNA PD1 expressing tumors (Cohort 3) | From date of allocation to death assessed up to approximately 36 months
  Time from allocation to death from any cause
PFS compared to PFS on prior line of therapy (pre-PFS) in patients with high mRNA PD1 expressing tumors (Cohort 3) | From date of allocation to disease progression or death from any cause,whichever came first, assessed up to approximately 36 months
  PFS on study treatment compared to PFS on prior line of therapy (pre-PFS).
ORR in patients with low mRNA PD1-expressing tumors (Cohorts 1 and 2) | Until objective tumor response, on average 10 months
  Proportion of patients with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
CBR in patients with low mRNA PD1 expressing tumors (Cohorts 1 and 2) | Until objective tumor response, on average 10 months
  Proportion of patients with a best overall response of CR, PR or an overall lesion response of Stable Disease (SD) or Non-PR/Non-progression disease (PD) lasting ≥ 24 weeks, based on local investigator´s assessment according to RECIST v1.1.
PFS in patients with low mRNA PD1 expressing tumors (Cohorts 1and 2) | From date of allocation to disease progression or death from any cause,whichever came first, assessed up to approximately 36 months
  Time from allocation to the first occurrence of disease progression, as determined locally by the investigator using RECIST v.1.1, or death from any cause, whichever occurs first.
DoR in patients with low mRNA PD1 expressing tumors (Cohorts 1and 2) | From date of allocation to disease progression or death from any cause,whichever came first, assessed up to approximately 36 months
  Time from the first occurrence of a documented objective response to disease progression, as determined locally by the investigator through use of RECIST v.1.1, or death from any cause, whichever occurs first
TtR in patients with low mRNA PD1 expressing tumors (Cohorts 1 and 2) | Until objective tumor response, on average 10 months
  Time from allocation to the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR.
OS in patients with low mRNA PD1 expressing tumors (Cohorts 1 and 2) | From date of allocation to death assessed up to approximately 36 months
  Time from allocation to death from any cause
PFS compared to PFS on prior line of therapy (pre-PFS) in patients with low mRNA PD1 expressing tumors (Cohorts 1 and 2) | From date of allocation to disease progression or death from any cause,whichever came first, assessed up to approximately 36 months
  PFS on study treatment compared to PFS on prior line of therapy (pre-PFS).
Incidence, seriousness, treatment-related and intensity of Treatment Emergent Adverse Events | During the whole treatment period (from baseline until patients' final treatment which is defined as the end of the Treatment Phase of the study, an average of 10 months
  Incidence, seriousness, treatment-related and intensity of Treatment Emergent Adverse Events (TEAEs) assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 5, including dose reductions, delays and treatment discontinuations.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo SOLTI, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Prat A, Paz-Ares L, Juan M, Felip E, Garralda E, Gonzalez B, Arance A, Martin-Liberal J, Gavila J, Lopez-Gonzalez A, Cejalvo JM, Izarzugaza Y, Amillano K, Corbacho JG, Saura C, Racca F, Hierro C, Sanfeliu E, Gonzalez X, Canes J, Villacampa G, Salvador F, Pascual T, Mesia R, Cervantes A, Tabernero J. SOLTI-1904 ACROPOLI TRIAL: efficacy of spartalizumab monotherapy across tumor-types expressing high levels of PD1 mRNA. Future Oncol. 2022 Oct 6. doi: 10.2217/fon-2022-0660. Online ahead of print. PMID 36200668